CLINICAL TRIAL: NCT05749068
Title: An Open-label Study to Evaluate the Use of the CapScan Intestinal Collection Device to Measure the Regional Metabolism of Sulfasalazine in the Digestive Tracts of Healthy Volunteers
Brief Title: Evaluation of the CapScan Device to Measure the Metabolism of Sulfasalazine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Envivo Bio Inc (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: EB-03; 1R21CA260665-01A1 (NIH)
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental (Experimental): Open label experimental arm
  Interventions: Device: CapScan intestinal sampling device

INTERVENTIONS:
Device: CapScan intestinal sampling device — CapScan is an intestinal collection device used to characterize the regional distribution of sulfasalazine, the metabolic breakdown products of sulfasalazine, and the gut microbiota in the digestive tracts of healthy volunteers.

SUMMARY:
Evaluation of the CapScan intestinal collection device in characterizing the metabolism of sulfasalazine in the digestive tracts of healthy volunteers.

DETAILED DESCRIPTION:
The objective is to evaluate the effectiveness of the CapScan intestinal collection device in characterizing the regional distribution of sulfasalazine, the metabolic breakdown products of sulfasalazine, and the gut microbiota in the digestive tracts of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older and 70 years of age or younger at the time of the first Screening Visit.

Physical Status Classification System 1 or 2. For women of childbearing potential, negative urine pregnancy test within 7 days of Screening Visit and agreement to remain abstinent (refrain from heterosexual intercourse) or use adequate contraception during the treatment period and for 14 days after the final dose of sulfasalazine.

Subject is fluent in English and understands the study protocol and informed consent and is willing and able to comply with study requirements and sign the informed consent form

Exclusion Criteria:

* • Known or suspected gastrointestinal obstructions, strictures or fistula

  * Known or suspected moderate to severe dysmotility, by the judgement of the principal investigator
  * Gastroparesis
  * A swallowing disorder
  * Known intolerance, reaction or hypersensitivity to sulfasalazine, its metabolites, sulfonamides, or salicylates
  * Urinary obstruction
  * Porphyria
  * Glucose-6-phosphate dehydrogenase deficiency
  * Known or suspected infection with severe acute respiratory syndrome, HIV, hepatitis B virus or hepatitis C virus
  * Pregnancy or planned pregnancy within 30 days from Screening Visit, or breast-feeding.
  * Use of concomitant medications, such as aspirin, antibiotics, laxatives and proton pump inhibitors that may interfere with the study in the judgement of the investigator.
  * Any form of active substance abuse or dependence (including drug or alcohol abuse), unstable medical or psychiatric disorder, or any chronic condition susceptible, in the opinion of the principal investigator, to interfere with the conduct of the study.
  * A clinical condition that, in the judgment of the principal investigator, could potentially pose a health risk to the subject while involved in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Silicon Valley Gastroenterology, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Regional Collection of Metabolites and Gut Microbiota
Description: Regional measurement of sulfasalazine in the intestinal lumen, the metabolic breakdown products of sulfasalazine and the gut microbiota in the digestive tracts of healthy volunteers.
Time Frame: 2 days
Measure: Number; unit: participants with sulfasalazine detected
Arm/Group | Experimental
Number analyzed (Participants) | 10
participants with sulfasalazine detected | 10

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT05749068/Prot_SAP_000.pdf